CLINICAL TRIAL: NCT00496587
Title: Phase II Safety and Efficacy Study of Capecitabine, Gemcitabine, and Bevacizumab in Combination for Patients With Metastatic or Unresectable Sarcomatoid Renal Cell Carcinoma
Brief Title: Capecitabine, Gemcitabine, and Bevacizumab in Combination for Patients With Sarcomatoid Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0433; NCI-2012-01511 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
Keywords: Genitourinary; Kidney Cancer; Sarcomatoid Renal Cell Carcinoma; Renal Cell Carcinoma; RCC; Sarcomatoid Carcinoma of the Kidney; Unresectable renal cell carcinoma; Capecitabine; Xeloda; Gemcitabine; Gemzar; Bevacizumab; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Avastin; Vascular Endothelial Growth Factor; VEGF
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Capecitabine; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine + Gemcitabine + Bevacizumab (Experimental): Capecitabine 800 mg/m^2 By Mouth Twice Daily On Days 1-21. Gemcitabine 900 mg/m^2 By Vein Over 30 Minutes on Days 1 and 15. Bevacizumab 10 mg/kg By Vein On Days 1 and 15.
  Interventions: Drug: Capecitabine; Drug: Gemcitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Capecitabine — 800 mg/m^2 By Mouth Twice Daily On Days 1-21.
  Other Names: Xeloda
Drug: Gemcitabine — 900 mg/m^2 By Vein Over 30 Minutes on Days 1 and 15.
  Other Names: Gemzar; Gemcitabine Hydrochloride
Drug: Bevacizumab — 10 mg/kg By Vein On Days 1 and 15.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF

SUMMARY:
The goal of this clinical research study is to learn if the combination of 3 drugs (gemcitabine, capecitabine, and bevacizumab) can help to control metastatic or unresectable renal cell carcinoma. The safety of this drug combination will also be tested.

DETAILED DESCRIPTION:
Gemcitabine and capecitabine are designed to disrupt the growth of cancer cells, which may cause cancer cells to start to die. Bevacizumab is a drug that binds to and inhibits Vascular Endothelial Growth Factor (VEGF), a blood-vessel stimulating agent with unusually high levels in kidney cancer.

If you are found to be eligible to take part in this study, you will receive gemcitabine, capecitabine, and bevacizumab on a 28 day cycle. Capecitabine will be taken by mouth (with food), twice daily, on Days 1-21. Gemcitabine will be given through a needle in your vein in your arm over 30 minutes on Days 1 and 15. Bevacizumab will be given through a needle in your vein in your arm on Days 1 and 15. It will be given over 120 minutes for Cycle 1 and over 60 minutes for all other cycles. Your doctor may decided to give you bevacizumab over 30 minutes if you tolerate the treatment well.

On the first day of each cycle, blood (about 2 teaspoons) and a urine will be collected before treatment for routine tests. You will also have blood drawn on Day 15 (about 2 teaspoons) for routine tests.

Every 8 weeks, you will have a CT scan of your chest, abdomen, and pelvis and a chest x-ray. You will be asked about any drugs that you are currently taking and you will have a complete physical exam. You will be asked about any side effects that you might have experienced since the last visit and your ability to perform daily activities will be evaluated. Repeat bone scans and MRI of the brain may be done if your doctor thinks it is necessary.

You will continue receiving treatment for a maximum of 12 months. However, if you are benefitting from treatment, you may be able to continue receiving it off study. You will be taken off study if the disease gets worse, if the side effects are intolerable, or if you develop another illness that prevents you from receiving the treatment.

This is an investigational study. Gemcitabine, capecitabine, and bevacizumab are all FDA approved and commercially available. Up to 40 participants may take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically demonstrated, metastatic or unresectable sarcomatoid carcinoma of the kidney, defined as the following: • A tumor biopsy (primary or metastasis) must show at least one focus of RCC (one of the recognized types); and, • A tumor biopsy (primary or metastasis) must have at least 10% of the sample showing sarcomatoid histology.
2. (# 1 cont'd) • Patients with primary tumor in place are eligible if there is any percentage of sarcomatoid dedifferentiation on a needle biopsy (primary or metastasis), and the radiographic appearance of the primary tumor on CT scan is typical of RCC. For these patients, due to the small tumor sample, it is not required to identify an area of typical RCC histology as long as the morphologic and immunostaining characteristics are consistent with RCC.
3. At least one site of measurable disease (may include primary tumor).
4. No prior cytotoxic chemotherapy. Any prior immunotherapy is permitted.
5. No prior bevacizumab treatment. Prior sorafenib or sunitinib is permitted.
6. Zubrod performance status 2 or better
7. Adequate organ and bone marrow function: • Absolute Neutrophil Count (ANC) >/= 1,500 • Platelets >/=100,000 • Total bilirubin </= 1.5 mg/dl • AST and ALT </= 3x upper limit normal • Creatinine clearance > 50 cc/min (measured or calculated by Cockcroft formula: Creatinine Clearance = [(140 - age) x wt (kg)]/[72 x creat (mg/dl)], for females x 0.85. Patients with creatinine clearance of 30-50 ml/min are eligible with an initial dose-reduction of capecitabine to the (-1) dose level.
8. Female patients of childbearing potential (last menses < 2 years) must have a negative blood pregnancy test within 7 days prior to starting treatment.
9. All patients must agree to practice adequate contraception if sexually active for the duration of the trial and for 2 months after discontinuation of the study drugs
10. Written informed consent.

Exclusion Criteria:

1. Patients with history of myocardial infarction, transient ischemic attack (TIA), stroke, pulmonary embolism, or history of deep vein thrombosis within the preceding 12 months.
2. Patients with major risk of bleeding, such as active brain metastases. Patients with controlled or small brain metastases will be eligible based on clinical assessment of the actual bleeding risk.
3. Patients with history of any major surgical procedure within the preceding 28 days.
4. Patients with baseline blood pressure >/= 140 systolic or >/= 90 diastolic.
5. Patients with nephrotic syndrome (proteinuria > 2 grams per 24 hours)
6. History of other malignancy, unless it is clinically non-threatening (such as non-melanoma skin cancer) or controlled for 2 years prior to study entry.
7. Prior treatment with gemcitabine, capecitabine, or any fluoropyrimidine.
8. Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-FU.
9. Any concurrent chemotherapy or radiotherapy.
10. Lack of physical integrity of the upper gastrointestinal tract, inability to swallow tablets or those who have malabsorption syndrome.
11. Clinically significant cardiac disease not well controlled with medication, such as symptomatic coronary artery disease, congestive heart failure, and cardiac arrhythmias.
12. Serious concurrent infections or other serious medical conditions, including uncontrolled diabetes.
13. Any serious non-healing wound, ulcer, or active bone fracture.
14. Any concurrent coumadin therapy. Patients who were previously on coumadin maintenance may switch to aspirin or low-molecular-weight heparin.
15. Patients who have had an organ allograft.
16. Unwillingness to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nizar M. Tannir, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 2, 2007 to February 24, 2012. All recruitment done at The University of Texas Cancer Center.
Groups:
- Capecitabine + Gemcitabine + Bevacizumab: Capecitabine 800 mg/m^2 orally twice daily Days 1-21; Gemcitabine 900 mg/m^2 intravenous (IV) Days 1 &15 and Bevacizumab 10 mg/kg IV Days 1 & 15.
Period: Overall Study
Arm/Group | Capecitabine + Gemcitabine + Bevacizumab
Started | 34
Completed | 3
Not Completed | 31
Not completed — Adverse Event | 2
Not completed — Progressive Disease | 24
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1
Not completed — Complications unrelated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 54 [38 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Event or disease-free survival given as progression free survival (PFS) which was defined as the length of time after primary treatment that the participant survives without disease progression. Evaluation of response will follow the Response Evaluation Criteria in Solid Tumors (RECIST) where progression is defined per RECIST criteria as an increase in disease of 20% or more in the sum of longest tumor diameters compared to baseline.
Time Frame: 12 months or until progression of disease
Population: One participant was excluded from survival analysis due to missing data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capecitabine + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 33
Months | 5.5 [3.4 to 7.7]

2. Primary Outcome: Time to Treatment Failure (TTF)
Description: Time to treatment failure, TTF, with failure defined as death or disease progression where progression is defined per RECIST criteria as an increase in disease of 20% or more in the sum of longest tumor diameters compared to baseline.
Time Frame: 12 months or until progression of disease
Population: Four participants were excluded from response analysis due to missing data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capecitabine + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 30
Months | 4.2 [2.4 to 6.0]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response defined as Complete Response + Partial Response, with response recorded from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Complete Response: The disappearance of all target lesions. Partial Response: >30% decrease in the sum of the longest diameter of target lesions, reference baseline sum longest diameter. Progressive Disease: At least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, or the appearance of one or more new lesions. Stable Disease: Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, reference smallest sum longest diameter since the treatment started.
Time Frame: 12 months or until progression of disease
Population: Four participants were excluded from response analysis due to missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine + Gemcitabine + Bevacizumab
Number analyzed (Participants) | 30
percentage of participants | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 28 day cycle up to one year with 12 cycles administered.
Arm/Group | Capecitabine + Gemcitabine + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 31/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine + Gemcitabine + Bevacizumab (N=34)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine + Gemcitabine + Bevacizumab (N=34)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8 (12)
Alkaline phosphatase (Investigations) | 10 (13)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (6) — including sneezing, nasal stuffiness, postnasal drip
Allergy/Immunology (Immune system disorders) | 5 (7)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 7 (9)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 19 (23)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 7 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 5 (7)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 4 (4)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3 (4)
Cardiac General-Other (Cardiac disorders) | 1 (1)
Cervical spine-range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (22)
Constitutional Symptoms (General disorders) | 1 (1)
Cough (General disorders) | 8 (17)
Creatinine (Investigations) | 12 (21)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 10 (26)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (24)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (2)
Dyspnea (Cardiac disorders) | 1 (1)
Dyspnea (shortness of breath) (Cardiac disorders) | 14 (23)
Edema: head and neck (Skin and subcutaneous tissue disorders) | 1 (1)
Edema: limb (Skin and subcutaneous tissue disorders) | 5 (5)
Endocrine (Endocrine disorders) | 5 (7)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 24 (69)
Fever (Blood and lymphatic system disorders) | 3 (4) — Fever (in absence neutropenia, where neutropenia is defined as ANC <1.0 x 10^9 per liter)
Gastrointestinal (Gastrointestinal disorders) | 5 (8)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 17 (45)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (3)
Hemoglobin (Blood and lymphatic system disorders) | 28 (54)
Hemoglobinuria (Blood and lymphatic system disorders) | 4 (4)
Hemorrhage, GU--Select (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 4 (7)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes/flushes (Reproductive system and breast disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (6)
Hypertension (Adult) (Endocrine disorders) | 2 (3)
Hypertension (Pediatric) (Endocrine disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Endocrine disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Joint (Musculoskeletal and connective tissue disorders) | 1 (3)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytes (Total WBC) (Blood and lymphatic system disorders) | 3 (8)
Lymphatics (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 8 (22)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Mood alteration (Psychiatric disorders) | 1 (1)
Mood alteration (Anxiety) (Psychiatric disorders) | 2 (2)
Mood alteration (Depression) (Psychiatric disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (clinical exam) (Oral Cavity) (Gastrointestinal disorders) | 5 (9)
Mucositis/stomatitis (functional/symptomatic) (Oral Cavity) (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (functional/symptomatic) (Stomach) (Gastrointestinal disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Extremity - lower) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 18 (40)
Neurology (Nervous system disorders) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 3 (7)
Neuropathy: sensory (Nervous system disorders) | 12 (29)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (5)
Obstruction, GI--Select (Small bowel NOS) (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 25 (95)
Pain--Select (Abdomen NOS) (Gastrointestinal disorders) | 4 (6)
Pain--Select (Back) (Musculoskeletal and connective tissue disorders) | 6 (10)
Pain--Select (Extremity-limb) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain--Select (Head/headache) (Nervous system disorders) | 3 (4)
Pain--Select (Neck) (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain--Select (Oral Cavity) (Gastrointestinal disorders) | 2 (2)
Pain--Select (Oral-gums) (Gastrointestinal disorders) | 1 (1)
Pain--Select (Pelvis) (Reproductive system and breast disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 5 (9)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (7)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 16 (29)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (4)
PTT (Partial Thromboplastin Time) (Investigations) | 1 (1)
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (18)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 19 (78)
Renal/Genitourinary (Renal and urinary disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Small/Large intestine (Gastrointestinal disorders) | 2 (3)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 9 (14)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (3)
Supraventricular and nodal arrhythmia--Select (Sinus tachycardia) (Cardiac disorders) | 2 (2)
Sweating (diaphoresis) (General disorders) | 5 (5)
Taste alteration (dysgeusia) (Nervous system disorders) | 7 (7)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 2 (3)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4 (5)
Urinary frequency/urgency (Renal and urinary disorders) | 3 (3)
Urine color change (Renal and urinary disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Voice changes/dysarthria (Nervous system disorders) | 3 (4) — e.g., hoarseness, loss or alteration in voice, laryngiti
Vomiting (Gastrointestinal disorders) | 10 (16)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes